CLINICAL TRIAL: NCT01556997
Title: Perindopril Amlodipine for the Treatment of Hypertension (PATH): A Multicenter, Randomized, Double-Blind, Parallel-Group Study Evaluating the Efficacy and Safety of a Fixed-Dose Combination of Perindopril Arginine Plus Amlodipine Besylate Versus Perindopril Erbumine and Amlodipine Besylate in Subjects With Essential Hypertension
Brief Title: Perindopril Amlodipine for the Treatment of Hypertension
Acronym: PATH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Symplmed Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X985400
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Results first posted 2015-08-25 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-08

CONDITIONS: Essential Hypertension
Keywords: Hypertension; Essential Hypertension
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Amlodipine; Perindopril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- XOMA 985 (Experimental): fixed-dose combination of perindopril arginine/amlodipine besylate(PERa/AMLb)
  Interventions: Drug: XOMA 985
- Amlodipine Besylate (AMLb) (Active Comparator)
  Interventions: Drug: Amlodipine Besylate
- Perindopril Erbumine (PERe) (Active Comparator)
  Interventions: Drug: Perindopril Erbumine

INTERVENTIONS:
Drug: XOMA 985 — PERa/AMLb capsule taken once daily by mouth for six weeks
  Arms: XOMA 985
Drug: Amlodipine Besylate — AMLb capsule taken once daily by mouth for six weeks
  Arms: Amlodipine Besylate (AMLb)
Drug: Perindopril Erbumine — PERe capsule taken once daily by mouth for six weeks
  Arms: Perindopril Erbumine (PERe)

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of a fixed-dose combination drug compared to two other drugs (monotherapies) in controlling hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension
* For female subjects, a negative serum pregnancy test
* Ability to provide written informed consent

Exclusion Criteria:

* Night shift workers whose work hours include midnight to 4:00 a.m.
* Secondary hypertension
* An arm size that precludes the use of the digital blood pressure monitor cuff (arm size > 42 cm)
* Renal dysfunction, severe renal impairment, bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, subjects with only 1 kidney, or post-renal transplant subjects
* Female subjects who are pregnant, planning to become pregnant
* History of malignancy within 5 years
* Primary aldosteronism
* Heart failure (NYHA functional class 3-4), hypertrophic obstructive cardiomyopathy, or hemodynamically relevant stenosis of the aortic or mitral valve
* Significant cardiac arrhythmias, MI, stroke, CABG, PTCA, unstable angina
* Known hypersensitivity to any component of the study drugs

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 837 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (48):
  - Huntsville, Alabama
  - Muscle Shoals, Alabama
  - Glendale, Arizona
  - Greenbrae, California
  - Los Angeles, California
  - Santa Ana, California
  - Denver, Colorado
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Palm Harbor, Florida
  - Port Orange, Florida
  - Marietta, Georgia
  - Gurnee, Illinois
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Louisville, Kentucky
  - Metairie, Louisiana
  - Auburn, Maine
  - Baltimore, Maryland
  - Olive Branch, Mississippi
  - Butte, Montana
  - Berlin, New Jersey
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Kettering, Ohio
  - Lyndhurst, Ohio
  - Marion, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - Austin, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Katy, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | XOMA 985 | Amlodipine Besylate (AMLb) | Perindopril Erbumine (PERe)
Started | 279 | 280 | 278
Completed | 253 | 252 | 246
Not Completed | 26 | 28 | 32
Not completed — Adverse Event | 10 | 12 | 12
Not completed — Lost to Follow-up | 6 | 6 | 4
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Withdrawal by Subject | 7 | 6 | 8
Not completed — Other | 2 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XOMA 985 | Amlodipine Besylate (AMLb) | Perindopril Erbumine (PERe) | Total
Number analyzed (Participants) | 279 | 280 | 278 | 837
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 261 | 262 | 254 | 777
  >=65 years | 18 | 18 | 24 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 130 | 143 | 407
  Male | 145 | 150 | 135 | 430
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 43 | 52 | 142
  Not Hispanic or Latino | 232 | 237 | 226 | 695
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 1 | 4
  Black or African American | 95 | 96 | 96 | 287
  White | 179 | 181 | 180 | 540
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 95 | 96 | 96 | 287
  Non-black | 184 | 184 | 182 | 550
Region of Enrollment [Number; unit: participants]
  United States | 279 | 280 | 278 | 837

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment in the Mean Seated Trough Cuff Diastolic Blood Pressure (DBP).
Time Frame: Day 0 to Day 42
Population: The Analysis Population for the Primary Outcome (Change from baseline to end of treatment in the mean seated trough cuff diastolic blood pressure (DBP)) consists of the Intent-to-treat population for the study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | XOMA 985 | Amlodipine Besylate (AMLb) | Perindopril Erbumine (PERe)
Number analyzed (Participants) | 271 | 275 | 274
mmHg | -15.7 (8.38) | -13.2 (8.33) | -9.5 (8.77)
Statistical Analysis 1: Comparison: XOMA 985 vs Amlodipine Besylate (AMLb) vs Perindopril Erbumine (PERe); Test type: Superiority or Other; p = 0.025, ANCOVA — The statistical model was an analysis of covariance model with treatment as the main effect and baseline DBP (<100 mmHg versus ≥100 mmHg), current type 2 diabetes status (yes versus no), and race (black versus non-black) as covariates

2. Secondary Outcome: Change From Baseline to End of Treatment in the Mean Seated Trough Cuff Systolic Blood Pressure (SBP).
Time Frame: Day 0 to Day 42
Population: The Analysis Population for the Secondary Outcome (Change from baseline to end of treatment in the mean seated trough cuff systolic blood pressure (SBP)) consists of the Intent-to-treat population for the study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | XOMA 985 | Amlodipine Besylate (AMLb) | Perindopril Erbumine (PERe)
Number analyzed (Participants) | 271 | 275 | 274
mmHg | -23.4 (13.86) | -19.6 (15.62) | -13.4 (14.66)
Statistical Analysis 1: Comparison: XOMA 985 vs Amlodipine Besylate (AMLb) vs Perindopril Erbumine (PERe); Test type: Superiority or Other; p = 0.025, ANCOVA — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: AE reporting began with Visit 1 and continued through 14 days after last dose, unless an unresolved AE was still being followed. At each evaluation, the Investigator determined whether any AEs occurred based on the criteria and definition of an AE or SAE. AEs may have been directly observed, elicited by Investigator, or volunteered by subjects.
Arm/Group | XOMA 985 | Amlodipine Besylate (AMLb) | Perindopril Erbumine (PERe)
Serious Adverse Events (participants affected / at risk) | 1/279 | 3/280 | 2/278
Other Adverse Events (participants affected / at risk) | 75/279 | 68/280 | 53/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XOMA 985 (N=279) | Amlodipine Besylate (AMLb) (N=280) | Perindopril Erbumine (PERe) (N=278)
Lip Swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XOMA 985 (N=279) | Amlodipine Besylate (AMLb) (N=280) | Perindopril Erbumine (PERe) (N=278)
Edema peripheral (General disorders) | 20 | 35 | 1
Fatigue (General disorders) | 5 | 2 | 4
Headache (Nervous system disorders) | 7 | 8 | 8
Dizziness (Nervous system disorders) | 7 | 3 | 4
Diarrhea (Gastrointestinal disorders) | 3 | 1 | 5
Nausea (Gastrointestinal disorders) | 2 | 2 | 4
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 8
Alanine amniotransferase increased (Investigations) | 0 | 0 | 4
Aspartate amniotransferase increased (Investigations) | 1 | 0 | 3
Blood potassium increased (Investigations) | 0 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Hematuria (Renal and urinary disorders) | 2 | 3 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No